# **African Surgical Outcomes Study in Paediatric patients (ASOS-Paeds)**

An African, international multi-centre fourteen-day evaluation of patient care and clinical outcomes for paediatric patients undergoing surgery

# STATISTICAL ANALYSIS PLAN VERSION 1.0

5 March 2025

# **Working Title:**

| An | evaluation | of intra-operative | severe | critical | events | in | ASOS-Paeds | (African | Surgical |
|---|---|---|---|---|---|---|---|---|---|
| Out | comes Stud | ly in Paediatric pa | tients): a | a 14-day | prospe | ctiv | e, observation | al cohort | study of |
| paed | diatric surgi | ical patients | | | | | | | |

**Emnet Tesfaye** 

First author, Co-investigator

Alexandra Torborg

Principal investigator

## **Contact details**

Principal investigator

## **Steering Committee for Study**

- 1. Alexandra Torborg MBChB FCA(SA), Discipline of Anaesthesiology and Critical Care Medicine, Nelson R. Mandela School of Medicine, University of KwaZulu-Natal, Durban, South Africa
- 2. Bruce Biccard MBChB FCA(SA) FFARCS(I) MMedSci PhD, Professor and Second Chair, Department of Anaesthesia and Perioperative Medicine, Groote Schuur Hospital and University of Cape Town, South Africa
- 3. Rupert Pearse MD(Res), Professor of Intensive Care Medicine, Queen Mary University of London, Royal London Hospital, London, E1 1BB, United Kingdom
- 4. Priyanka Naidu MBChB, Department of Research, Education, and Innovation, Operation Smile, Virginia Beach, Virginia, USA, Centre for Global Surgery, Department of Global Health, Stellenbosch University, Tygerberg, South Africa.
- 5. Hyla Kluyts DMed (Anaest), Department of Anaesthesiology, Sefako Makgatho Health Sciences University, South Africa
- 6. Mary T. Nabukenya MMED, FCA(ECSA), Lecturer, Makerere University College of Health Sciences, Paediatric anaesthesiologist, Mulago National Referral Hospital, Kampala, Uganda
- Adesoji O Ademuyiwa, FACS, Professor of Surgery (Paediatric and Surgical Epidemiology), Department of Surgery, College of Medicine, University of Lagos and Lagos University Teaching Hospital, Lagos, Nigeria

## Writing group for Anaesthesia Critical Incidents Paper

First Author Emnet Tesfaye

Co-Authors Alexandra Torborg Gwen Arendse Bruce Biccard

# **Table of Contents**

| Introduction and rationale for the "severe critical events" analysis | 4 |
|---|---|
| Aims and objectives of the "severe critical incidents" analysis | 5 |
| Aims | |
| Objectives of the study | 5 |
| Statistical Analysis Plan | 7 |
| A) Data Validation | 7 |
| B) Statistical tests | 7 |
| C) Primary objective | 7 |
| D) Secondary objectives | 8 |
| Tables | 9 |
| Table 1. Description of cohort including patient, surgical, anaesthesia and facility characteristics | 9 |
| Table 2: The categories and types of intra-operative severe critical events | 11 |
| Table 3. Univariable and multivariable analysis of preoperative factors associated with intra-operative | 'e |
| severe critical events | 12 |
| Table S1: Intra-operative severe critical events by facility and anaesthesia provider | 14 |
| References | 16 |

## Introduction and rationale for the "severe critical events" analysis

Universal Health Coverage aims to guarantee access to needed health care services for all people without financial burden, which includes surgical service delivery. (1) The World Health Assembly resolution EB152(3), stated "integrated Emergency Critical Operative Care for universal health care (ECO-UHC) and protection from health emergencies" should be part of global health improvement interventions. It advocates for the delivery of quality health care for acutely ill people. This includes early access and intervention for general acute childcare including operative care. This is particularly important in low and middle income countries because the proportion of child population is estimated to be half of the total population. (2)

Paediatric mortality after surgical procedures continues to be high. One study reported a mortality of 12%, with oesophageal atresia accounting for 72% and jejunoileal atresia for 35%. (3) The human resources available for paediatric surgery are limited, with a low number of paediatric surgeons and paediatric anaesthesiologists compared to the burden of the paediatric surgical population. The result is that in many places non-specialists and even other non-physician professionals might be solely responsible for peri-operative care. (4,) (5) This can result in excess intra-operative critical events. Critical events are however, inadequately investigated in Africa. The existing data are derived from registries which are often incomplete and may not target critical events.

Intraoperative critical events can have multiple risk factors and contribute to anaesthesia related complications. The incidence ranges from 2.32% to 11.7% and shows significant variability among different settings. The largest intraoperative critical event study in Europe showed a high number of intraoperative severe critical events (5.2%) with significant variability between hospitals. Respiratory critical events were the most common (3.1%) followed by cardiovascular instability (1.9%). The immediate poor outcome was 5.4%. (6)

There are specific considerations that should be sought in Paediatric population aesthesia related critical events. These may include the choice of drug and their response. Additionally, the anaesthesia related adverse effects may have long term sequelae for children. As a result, studying those critical events will help to identify the factors related and final outcomes which will help in standardizing the care. It will also be a base to advocate for intraoperative care.

### Reported incidences from high income countries

Studies from Europe reported incidences ranging from 0.14% for serious adverse events to 3.4% for critical incidents. (7) Similarly a study done by Cohen et al showed a severe anaesthesia critical event rate of 1.4 per 1000. The commonest events were respiratory followed by cardiac. (8) A large international multicentric cohort study covering North America, Oceania and Europe reported an incidence of 24% for intraoperative adverse events. (9)

## Reported incidences from low- and middle-income countries

The reported incidences for critical events vary across low and middle-income countries (LMICs). A South Korean study reported a 0.4% incidence of paediatric anaesthesia related critical incidents, with respiratory events been the commonest (55% of the cases), (10) compared to an Indian study which reported a 12% incidence, predominated by respiratory complications. (11) Generally, LMICs may carry at least double the burden of intraoperative critical events to high-income countries, although the risk should be similar to that of HICs. These excess events should be preventable. (12)

## *Types of complications*

Respiratory related complications are most commonly reported, followed by cardiovascular events.

### Risks associated with complications

The following patient and surgical risk factors have been shown to contribute to intraoperative critical events: age <1 year, ASA physical status III and IV, urgency of the surgical procedure, and preexisting comorbidities. The level of training of the anaesthesia providers and the number of years of experience, as well as the type of anaesthesia and surgery done are potentially important risk factors. (13)

## Study rationale

African Surgical Outcomes Study in Paediatric patients (ASOS-Paeds) determined the incidence of in-hospital postoperative complications up to 30 days after surgery in paediatric surgical patients across different hospitals in Africa. This study will evaluate the intra-operative critical incidents reported in ASOS-Paeds. It is hoped that these findings will contribute to improving perioperative care for paediatric surgical patients in Africa.

## Aims and objectives of the "severe critical incidents" analysis

#### Aims

The aims of this study are to describe the incidence of intraoperative severe critical events, the types of severe critical events, and risk factors independently associated with severe critical events.

## Objectives of the study

Primary objective

1. To describe the incidence of intra-operative severe critical events in paediatric surgical patients in Africa

## Secondary objectives

- 1. To describe the categories and types of severe critical events
- 2. To identify risk factors independently associated with severe critical events

## Sensitivity analyses

- 1. Two sensitivity analyses will be conducted:
  - a. The sensitivity analyses of elective surgical patients, and emergency surgical patients, and
  - b. A sensitivity analysis excluding the two countries providing more than 10% of the patients to the dataset (Egypt and South Africa)

## Statistical Analysis Plan

## A) Data Validation

- Report on the number of incomplete data points
- Report on primary outcome data
  - o % missing data for incidence of severe critical events
- Provide STROBE diagram of recruited patients

### B) Statistical tests

- Categorical variables will be described as number and proportions (percentage) and will be compared using appropriate Chi-squared or Fisher's exact tests.
- Continuous variables will be calculated and reported as mean and standard deviation (SD) if normally distributed, or median and inter-quartile range (IQR) if not normally distributed.
- Comparisons of continuous variables between groups will be performed using t-tests, one-way ANOVA or equivalent non-parametric tests as appropriate.
- If < 5% of data are missing for the primary outcomes, a complete case analysis will be conducted
- A p-value of less than 0.05 will be considered statistically significant for all analyses
- Generalized mixed effects model analysis will be performed for exploration of candidate variables for prediction of risks for the primary outcome i.e. incidence of severe critical events
  - o Further description to follow in the section discussing risk prediction
- Sensitivity analyses will be conducted.

## C) Primary objective

1. To describe the incidence of intra-operative severe critical events in paediatric surgical patients in Africa

This will be presented as number (n/N), percentage (%)

The cohort will be described according to the variables (Table 1)

- Age, ASA PS, sex
- Comorbidities
- Describe the Hospital, Surgery and Anaesthesia information
  - Hospital level
  - Urgency of surgery (elective, emergency)
  - o Severity of surgery (minor, intermediate, severe),
  - Indication for surgery
  - o Type of surgery
  - Intraoperative factors
  - Most senior anaesthetist
  - Most senior surgeon

#### o Time of induction

## D) Secondary objectives

- 1. To describe the categories and type of intra-operative severe critical events
- Outcome definitions are defined in the study protocol
  - The categories of severe critical events will be presented as airway, respiratory, cardiovascular, metabolic, and other severe critical events categories (Table 2) using % to indicate the incidence (number of patients with severe critical events divided by the number of patients) and 95% confidence intervals.
  - o To describe the types of severe critical events within each category
  - The categories and types of severe critical events will also be presented by the level of facility, and the level of the anesthesia providers (Table S1)
- 2. To identify risk factors independently associated with severe critical events
- All variables will be entered into the model, unless there are less than 10 events per variable. If this is the case, risk factors with a p value ≤ 0.05 for severe critical events identified by univariate analysis will be entered into the model. (Table 3) The reference category for the surgical discipline will be decided by the surgical discipline with the lowest incidence of severe critical events
  - Results will be presented as unadjusted and adjusted odds ratios (ORs) with 95% confidence intervals (CI's).

Analyses will be conducted using Statistical Package for the Social Sciences (SPSS) version 30 (SPSS Inc., Chicago, IL, USA) and R: A language and environment for statistical computing. Vienna, Austria: R Foundation for Statistical Computing (2024) using Studio: Integrated Development Environment for R. Boston, MA: RStudio, Inc. (2024).

# Tables

Table 1. Description of cohort including patient, surgical, anaesthesia and facility characteristics

| | | All patients (n= ) | Patients with severe critical events (n=) | Patients without severe critical events (n=) |
|---|---|---|---|---|
| | | n/N (%) | n/N (%) | n/N (%) |
| Age | Mean (SD) | | | |
| | Median (IQR) | | | |
| Sex | | | | |
| Mal | | | | |
| Fem | | | | |
| | tegories | | | |
| | 3 days | | | |
| | lays to < 1 yr | | | |
| | < 4 yr | | | |
| | < 13 yr | | | |
| | o <18 yr | | | |
| ASA PS | S | | | |
| I | | | | |
| II | | | | |
| III | | | | |
| IV- | V | | | |
| Urgenc | y of surgery | | | |
| Rou | ıtine | | | |
| Eme | ergency | | | |
| Severit | y of surgery | | | |
| Min | ior | | | |
| Inte | rmediate | | | |
| Maj | or | | | |
| Primar | y indication for | | | |
| surgery | 7 | | | |
| Nor | n-communicable | | | |
| dise | ease | | | |
| Infe | ective | | | |
| Trai | uma | | | |
| Con | genital | | | |
| Hospita | <u> </u> | | | |
| Firs | | | | |
| Sec | ond | | | |
| Thi | | | | |
| | enior anaesthetist | | | |

| Specialist |
|---------------------------|
| Non-specialist physician |
| Nurse |
| Non-physician |
| Most senior surgeon |
| Specialist |
| Non-specialist physician |
| Nurse |
| Non-physician |
| Type of surgery |
| Orthopaedic |
| Cardiac |
| ENT |
| Gynaecological |
| Hepatobiliary |
| Kidney/urological |
| Gastrointestinal |
| Thoracic |
| Ophthalmology |
| Maxillo-facial/ dental |
| Plastic/cutaneous |
| Neurosurgery |
| Burns |
| Comorbidities |
| Cardiac disease |
| Chronic respiratory |
| disease |
| Neurological disorder |
| HIV/AIDS |
| Cancer |
| Current respiratory tract |
| infection |
| Intraoperative factors |
| Duration |
| Surgical checklist used |
| Time |
| Daytime |
| After hours |

Table 2: The categories and types of intra-operative severe critical events

| | Overall | Incidence |
|------------------------------------|---------|------------|
| | n/N (%) | % (95% CI) |
| Categories of anaesthetic severe | | |
| critical incidents | | |
| Any | | |
| Any Airway/respiratory | | |
| Any CVS | | |
| Any Other | | |
| Types of severe critical events by | | |
| category | | |
| Airway/respiratory | | |
| Difficult BMV | | |
| Difficult Intubation | | |
| Failed Intubation | | |
| Laryngospasm | | |
| Bronchospasm | | |
| Aspiration | | |
| Severe Hypoxia | | |
| CVS | | |
| Bradycardia | | |
| Cardiovascular instability | | |
| Cardiac Arrest | | |
| Metabolic | | |
| Temp < 36 | | |
| Low Glucose | | |
| Other | | |
| Anaphylaxis | | |
| Drug error | | |
| Death | | |
| Yes | | |
| No | | |

Table 3. Univariable and multivariable analysis of preoperative factors associated with intra-operative severe critical events

| | Univariable | | Multivariable | |
|------------------------|-------------|---------|---------------|---------|
| | OR (95% CI) | p-value | OR (95% CI) | p-value |
| Age (per 1 year) | | | | |
| Sex | | | | |
| Male | | | | |
| Female | Reference | | | |
| ASA PS | | | | |
| I | Reference | | | |
| II | | | | |
| III | | | | |
| IV-V | | | | |
| Urgency of surgery | | | | |
| Routine | Reference | | | |
| Emergency | | | | |
| Severity of surgery | | | | |
| Minor | Reference | | | |
| Intermediate | | | | |
| Major | | | | |
| Primary indication for | | | | |
| surgery | | | | |
| Non-communicable | Reference | | | |
| disease | | | | |
| Infective | | | | |
| Trauma | | | | |
| Congenital | | | | |
| Hospital level | | | | |
| First | | | | |
| Second | | | | |
| Third | Reference | | | |
| Most senior surgeon | | | | |
| Specialist | Reference | | | |
| Non-specialist | | | | |
| physician | | | | |
| Nurse | | | | |
| Non-physician | | | | |
| Most senior | | | | |
| anaesthetist | | | | |
| Specialist | Reference | | | |

| NT ' 1' 4 | |
|------------------------|-----------|
| Non-specialist | |
| physician | |
| Nurse | |
| Non-physician | |
| Type of surgery | |
| Orthopaedic | |
| Cardiac | |
| ENT | |
| Gynaecological | |
| Hepatobiliary | |
| Kidney/urological | |
| Gastrointestinal | |
| Thoracic | |
| Ophthalmology | |
| Maxillo-facial/ | |
| dental | |
| Plastic/cutaneous | |
| Neurosurgery | |
| Burns | |
| Comorbidities | |
| Cardiac disease | |
| Chronic respiratory | |
| disease | |
| Neurological | |
| disorder | |
| HIV/AIDS | |
| Cancer | |
| Current respiratory | |
| tract infection | |
| Intraoperative factors | |
| Duration | |
| Surgical checklist | Reference |
| used | |
| Surgical checklist | |
| not used | |
| Time | |
| Daytime | Reference |
| After hours | |

Table S1: Intra-operative severe critical events by facility and anaesthesia provider

| | Hospital level | | | Most senior anaesthetist | | | |
|---|---|---|---|---|---|---|---|
| | District | Regional | Tertiary | Specialist | specialist | Nurse | Non-<br>physician |
| | | | | | physician | | |
| Categories of anaesthetic severe critical incidents | | | | | | | |
| Any | | | | | | | |
| Any Airway/respiratory | | | | | | | |
| Any CVS | | | | | | | |
| Any Other | | | | | | | |
| Types of severe critical | | | | | | | |
| events by category | | | | | | | |
| Airway/respiratory | | | | | | | |
| Difficult BMV | | | | | | | |
| Difficult Intubation | | | | | | | |
| Failed Intubation | | | | | | | |
| Laryngospasm | | | | | | | |
| Bronchospasm | | | | | | | |
| Aspiration | | | | | | | |
| Severe Hypoxia | | | | | | | |
| CVS | | | | | | | |
| Bradycardia | | | | | | | |
| Cardiovascular | | | | | | | |
| instability | | | | | | | |

| Cardiac Arrest |
|----------------|
| Metabolic |
| Temp < 36 |
| Low Glucose |
| Other |
| Anaphylaxis |
| Drug error |
| Death |
| Yes |
| No |

### References

- 1. Stuckler D, Feigl A, Basu S, McKee M. The political economy of universal health coverage. Background paper for the global symposium on health systems research. 2010;
- 2. The World Health Assembly resolution on integrated emergency, critical, and operative care for universal health coverage and protection from health emergencies: a golden opportunity to attenuate the global burden of acute and critical illness. Intensive Care Medicine. 2023;49(10):1223–5.
- 3. Livingston MH, DCruz J, Pemberton J, Ozgediz D, Poenaru D. Mortality of pediatric surgical conditions in low and middle income countries in Africa. Journal of pediatric surgery. 2015;50(5):760–4.
- 4. Chirdan LB, Ameh EA, Abantanga FA, Sidler D, Elhalaby EA. Challenges of training and delivery of pediatric surgical services in Africa. Journal of pediatric surgery. 2010;45(3):610–8.
- 5. Tyson AF, Msiska N, Kiser M, Samuel JC, Mclean S, Varela C, et al. Delivery of operative pediatric surgical care by physicians and non-physician clinicians in Malawi. International Journal of Surgery. 2014;12(5):509–15.
- 6. Habre W, Disma N, Virag K, Becke K, Hansen TG, Jöhr M, et al. Incidence of severe critical events in paediatric anaesthesia (APRICOT): a prospective multicentre observational study in 261 hospitals in Europe. The Lancet Respiratory Medicine. 2017;5(5):412–25.
- 7. De Graaff JC, Sarfo M, Van Wolfswinkel L, van der Werff DB, Schouten AN. Anesthesia-related critical incidents in the perioperative period in children; a proposal for an anesthesia-related reporting system for critical incidents in children. Pediatric Anesthesia. 2015;25(6):621–9.
- 8. Kurth CD, Tyler D, Heitmiller E, Tosone SR, Martin L, Deshpande JK. National pediatric anesthesia safety quality improvement program in the United States. Anesthesia & Analgesia. 2014;119(1):112–21.
- 9. Dell-Kuster S, Gomes NV, Gawria L, Aghlmandi S, Aduse-Poku M, Bissett I, et al. Prospective validation of classification of intraoperative adverse events (ClassIntra): international, multicentre cohort study. Bmj. 2020;370.
- 10. Lee J, Kim E, Song I, Kim E, Kim H, Kim C, et al. Critical incidents, including cardiac arrest, associated with pediatric anesthesia at a tertiary teaching children's hospital. Pediatric Anesthesia. 2016;26(4):409–17.
- 11. Mittal A, Agarwal M. Analysis of critical incidents in pediatric anaesthesia-a clinical study. Journal of Advanced Medical and Dental Sciences Research. 2017;5(1):131.

- 12. Cronje L. A review of paediatric anaesthetic-related mortality, serious adverse events and critical incidents. Southern African Journal of Anaesthesia and Analgesia. 2015;21(6):5–11.
- 13. von Ungern-Sternberg BS, Boda K, Chambers NA, Rebmann C, Johnson C, Sly PD, et al. Risk assessment for respiratory complications in paediatric anaesthesia: a prospective cohort study. The Lancet. 2010;376(9743):773–83.